CLINICAL TRIAL: NCT03239834
Title: Clinical Evaluation of the OncAlert RAPID; Impact on Decision-Making
Brief Title: Clinical Evaluation of the OncAlert RAPID in Subjects Presenting for Evaluation and/or Initial Biopsy; Impact on Decision-Making
Status: Completed | Type: Observational
Sponsor: Vigilant Biosciences, Inc. (Industry)
Collaborators: Pearl Pathways (Unknown)
Responsible Party: Sponsor
Other Study IDs: VIG-001
Record Dates: First submitted 2017-06-19; First posted 2017-08-04 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Palatal Neoplasms; Lip Neoplasm; Gingival Neoplasms; Leukoplakia, Oral; Tongue Neoplasms; Oropharyngeal Neoplasms; Oral Ulcer
MeSH Terms: conditions — Palatal Neoplasms; Lip Neoplasms; Gingival Neoplasms; Leukoplakia, Oral; Tongue Neoplasms; Oropharyngeal Neoplasms; Oral Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- OncAlert RAPID test in oral cavity biopsy patients.: Patients at an intermediate and high level of clinical risk for HNSCC and scheduled for initial and immediate incisional diagnostic biopsy of their Oral Cavity.
  Interventions: Device: OncAlert
- OncAlert RAPID test in oropharyngeal biopsy patients.: Patients at an intermediate to high level of clinical risk for HNSCC and scheduled for initial and immediate incisional diagnostic biopsy of their Oropharnyx
  Interventions: Device: OncAlert
- OncAlert RAPID test in clinical decision to biopsy.: Patients at a lower level of clinical risk for HNSCC and not scheduled for an immediate biopsy. Patients will be offered medical management and have an initial RAPID test. All patients will return within 1-3 months for follow-up test and a possible biopsy if clinically indicated.
  Interventions: Device: OncAlert

INTERVENTIONS:
Device: OncAlert — A noninvasive point of care salivary rinse test performed as 1) a one-time test for patients presenting with suspicion of OPMD and scheduled for biopsy and 2) a multi-administered test for patients presenting with suspicious lesions not scheduled for biopsy.

SUMMARY:
Objectives Validate the OncAlert® RAPID Test by demonstrating that NPV > (1 -prevalence).

Evaluate the independent and associated contribution of readily available clinical variables including age, race, gender, HPV status, socioeconomic level, tobacco, and alcohol use with the biopsy and test results.

Evaluate OncAlert® RAPID Test results in patients without immediate biopsy, both at baseline and scheduled follow-up visit (approximately 1-3 months±14 days), to assess impact on outcome.

Planned Number of Subjects A total enrollment of up to 1000 individuals is projected with 600 as the minimum accrued. Patients in the primary cohort (1a and 1b) will be followed until pathology of clinically directed incisional / diagnostic biopsy pathology report is received.

Up to 200 'non-biopsy subjects' will be followed during a 1-3 month ±14 days clinic visit.

Patient Population

Cohorts 1a and 1b:

Subjects with a clinical suspicion of oral potentially malignant disorders, oral or oropharyngeal cancer, or both based in part on clinical examination, symptoms, clinical history, suspicious lesion(s) in mouth without history of a prior positive biopsy. Even if the suspicion is low for cancer or precancer, the patient is eligible if a biopsy is performed, in part, to rule this out. For example, if a subject has findings on imaging, or worrisome localizing symptoms in the oral cavity or oropharynx, they would be eligible. In addition, subjects with papillomas or other findings where there is a low level of concern, but cancer is still in the differential, are also eligible.

* Cohort 1a: oral cavity
* Cohort 1b: oropharynx

Cohort 2:

Subjects are enrolled with a clinical suspicion of oral potentially malignant disorders, oral or oropharyngeal cancer, or both based in part on clinical examination, symptoms, clinical history, suspicious lesion(s) in mouth without history of a prior positive biopsy; however, based on clinical impression and or patient related issues no immediate biopsy is obtained.

Screen Fail Rate: A 20% Screen Fail Rate is anticipated.

Investigational Product Name: OncAlert Oral Cancer RAPID Test (OncAlert RAPID)

Methodology Overview

Prospectively collect 5cc of normal saline after a combination of swish, gargle and spit into the provided collection specimen cup. Specimens will be collected at baseline (time of biopsy) as per standard practice at each site. The OncAlert RAPID Test cassette is inserted into the specimen cup and read directly from the cassette in 10 minutes. In addition, comprehensive clinical - pathology and patient demographic features including age, gender, race, ethnicity, and all pathology biopsy results will be collected. Any pertinent additional clinical data including HPV status, socioeconomic status, smoking, drinking history, and pertinent features related to oral health will be obtained. A central pathology review for all biopsy results will be performed and incorporated into the final analyses.

DETAILED DESCRIPTION:
Overview

The OncAlert Oral Cancer RAPID Test (OncAlert RAPID) is a qualitative point-of-care lateral flow assay to aid in the decision to biopsy in patients with clinical features associated with oral potentially malignant disorders and or oral/oropharyngeal cancer (i.e. head and neck squamous cell carcinoma).

Proposed Intended Use Statement

The device measures soluble CD44 and total protein in saliva samples collected in saline. The test is an adjunct to the biopsy decision process, and not intended as a screening or stand-alone diagnostic assay. To be used in adults 23 years and older. Not intended for use in pregnant women.

STUDY OBJECTIVES

The principal objectives of this study are to:

* Validate the OncAlert RAPID Test, with an NPV ≥ (1-prevalence),
* Evaluate OncAlert RAPID Test results in patients without immediate biopsy, both at baseline and scheduled follow-up visit (approximately 1-3 months), to assess impact on outcome,
* Evaluate the independent and associated contribution of readily available clinical variables including age, race, gender, HPV status, socioeconomic level, tobacco, and alcohol use with the biopsy and test results.

STUDY OVERVIEW

Study Approach

Prospectively collect 5cc of normal saline after a combination of swish, gargle and spit into the provided collection specimen cup. 1cc will be removed and sequestered for subsequent downstream analyses (Section 7). Specimens will be collected at baseline (time of biopsy) as per standard practice at each site. The OncAlert RAPID Test cassette is inserted into the specimen cup and read directly from the cassette in 10 minutes. In addition, acquire comprehensive clinical - pathology and patient demographic features including age, gender, race, ethnicity, and all pathology biopsy results. Also, obtain any pertinent additional clinical data including HPV status, socioeconomic status, smoking, drinking history, and pertinent features related to oral health. It is presumed that some patients within the current biopsy protocol will undergo treatment as a result of the biopsy diagnosis. The clinical-pathology data, when accessible, for these patients will be collected for subsequent secondary analyses. A central pathology review for all biopsy results will be performed and incorporated into the final analyses.

Study Duration

For Cohorts 1a and 1b patients, the pathology results of clinically directed incisional / diagnostic biopsy will be followed until finalized and received.

Cohort 2 patients not having an initial incisional / diagnostic biopsy at the initial visit will have an additional OncAlert® RAPID test performed within 1 -3 months±14 days (or as defined by standard of care (SOC)after the initial visit.)

The study will conclude after all data is collected and analyzed. This could vary from 12 to 36 months or more depending on accrual rates at the open sites and other factors.

ELIGIBILITY:
Inclusion Criteria:

* 23 years of age or older
* A clinical suspicion of oral potentially malignant disorders, oral or oropharyngeal cancer, or both based in part on clinical examination, symptoms, clinical history, suspicious lesion(s) in mouth without history of a prior positive biopsy.
* The subject must be able to comprehend and sign an approved Informed Consent Form and other applicable study documents.
* Patients are eligible regardless of race, gender, and ethnicity

Exclusion Criteria:

* Prior history and/or diagnosis of any HN cancer/HNSCC of the oral cavity, oropharynx, or hypopharynx including nasopharyngeal carcinoma.
* Prior treatment of HN cancer / HNSCC of the oral cavity, oropharynx, or hypopharynx including nasopharyngeal carcinoma.
* Prior history of a positive biopsy of the oral cavity or oropharynx.
* Planned excisional biopsy for a pathology diagnosis of HNSCC
* Clinical presentation without localizing findings
* Prior history of a salivary gland tumor
* Current and or prior diagnosis of cancer (note: other than basal and squamous cell carcinoma of the skin) within the past 5 years.
* Pregnant

Min Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the current study cohort,we anticipate working with 20 or more institutions to obtain oral rinse saliva samples from up to 1000patients (most patients scheduled for biopsyof the oral cavity or oropharynx and not more than 200 non-biopsy patients) from different geographic regions.
  The study population will be representative of adults at least 23 years of age who have been diagnosed as described in inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 893 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Association of RAPID results with oral cavity / oropharyngeal biopsy. | 18 months
  The likelihood of a positive biopsy was determined when either the presence of a CD44 band or Total Protein above a specific gradient were positive.
Association of RAPID results with the clinical decision process for avoiding an immediate biopsy. | 18 months
  Evaluate OncAlert RAPID results in patients without immediate biopsy, both at baseline and repeat results at scheduled follow-up visit (approximately 1-3 months). If biopsy performed associate RAPID positive vs. negative results with biopsy outcome. If not biopsy is performed, compare results with clinical decision for not to biopsy.

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Dr. Joel Epstein, Beverly Hills, California
  - Biosolutions Clinical Research Center, La Mesa, California
  - Loma Linda School of Dentistry, Loma Linda, California
  - Tower ENT, based at Cedars Sinai Medical Center, Los Angeles, California
  - Sacramento ENT, Roseville, California
  - Sacramento ENT, Sacramento, California
  - UConn Dental Medicine, Farmington, Connecticut
  - University of Miami Health Systems, Miami, Florida
  - ENT of South Florida Plantation, Plantation, Florida
  - ENT of South Florida Port St. Lucie, Port Saint Lucie, Florida
  - Asclepes Research, Weeki Wachee, Florida
  - Chicago ENT, Chicago, Illinois
  - Heartland Medical Research, Clive, Iowa
  - University of Maryland, Baltimore, Maryland
  - Tufts University, Boston, Massachusetts
  - Boston University Dental School, Boston, Massachusetts
  - UMKC School of Dentistry, Kansas City, Missouri
  - Duke Head and Neck Surgery & Communication Services, Durham, North Carolina
  - Eastern Carolina University School of Dental Medicine, Greenville, North Carolina
  - Piedmont Ear, Nose and Throat Associates, Winston-Salem, North Carolina
  - Specialty Physician Associates, Bethlehem, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis, Tennessee
  - Fort Worth ENT, Fort Worth, Texas
  - Berkson Medical, LLC, Mansfield, Texas
  - Chrysalis Clinical Research, St. George, Utah

IPD SHARING:
Plan to Share IPD: No